## Effect of Injectable Platelet-Rich Fibrin (i-PRF) in Initial Treatment of Chronic

## **Periodontitis**

- NCT04178590
- 26 April, 2020

## Statistical analysis

Statistical Package for Social Science (SPSS software package, version 26.0; SPSS Inc., Chicago, IL, USA) was used for all the data analyses. For numerical data, mean values, medians, standard deviations (SD) and ranges were used for description. The distributions of all outcome values were examined using the Kolmogorov–Smirnov normality test and depending on the distribution, measurements at baseline and at each follow-up between two treatment groups were compared using paired Student's t-test or Wilcoxon signed-rank test. Comparisons within each treatment group for all the measurements were done by repeated measures ANOVA with Bonferroni correction or Friedman and Wilcoxon signed-rank test. Univariate and multivariate logistic regression models were used to assess the predictors of difference between treatment groups. Univariate and multivariate linear regression models were for the predictors of primary outcome (CAL) at 6 months. The differences were considered as significant when the p value was <0.05. Study power was calculated using DSS Research, for primary outcome (CAL) at 6 months and it was above 90%.